CLINICAL TRIAL: NCT01995864
Title: A Pilot Multi-center Randomized Controlled Trial of Critical Time Intervention - Task Shifting (CTI-TS) Versus Usual Care for People With Psychotic Disorders
Brief Title: Critical Time Intervention-Task Shifting: Randomized Controlled Trial
Acronym: CTI-TS RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ezra S. Susser, MD, DrPH, Professor of Epidemiology and Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAI1845; U19MH095718 (NIH)
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia; Psychotic Disorder
Keywords: Schizophrenia and Disorders with Psychotic Features; Community Psychiatry
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTI-TS (Experimental): CTI-TS is a time-limited, 9-month long intervention, provided at the critical time when a person is first offered services at a mental health clinic, or, at the similarly critical time when a person first seeks to reconnect with a mental health clinic after a long lapse.
  Interventions: Behavioral: CTI-TS
- Usual Care (No Intervention): The Usual Care group will receive mental health services as provided by the local mental health services clinic.

INTERVENTIONS:
Behavioral: CTI-TS — The following briefly describes the three phases of CTI-TS:
  Phase 1: Initiation: The client and CTI-TS team formulate a treatment plan that focuses on selected areas identified as crucial for strengthening stability and facilitating the assimilation of the individual into community living.
  Phase 2: The Try-Out phase is devoted to testing and adjusting the support systems that have been established in the community.
  Phase 3: The final phase, Transfer of Care, is devoted to making any necessary improvements in the network of supports of the individual.
  Other Names: CTI-TS (Critical Time Intervention-Task Shifting)
  Arms: CTI-TS

SUMMARY:
The study represents the research component of a broader initiative entitled "RedeAmericas". RedeAmericas (RA) is a collaborative effort of investigators from six cities across Latin America (Buenos Aires, Cordoba, Medellin, Neuquen, Rio de Janeiro, and Santiago) and Columbia University in New York.

This is a pilot Randomized Controlled Trial (RCT) of Critical Time Intervention-Task Shifting (CTI-TS). It is designed to address a fundamental gap in the services offered by mental health clinics. These clinics are the primary locale for outpatient treatment of individuals with severe mental disorders in the urban areas of Latin America, and they offer some basic and important clinical care such as pharmacologic treatment onsite. Generally these clinics also have a major limitation; they have inadequate resources and training for the provision of in vivo community-based services, that is, services delivered outside of the clinic facility in homes or elsewhere in the community. In most urban areas, they also have weak links to primary health care and are not easily accessible to much of the population.

CTI-TS, is a task shifting intervention that at the service user level provides support for better community living and promotes social integration, and at the system level strengthens the connections between mental health and primary care clinics. CTI-TS is a time-limited 9-month intervention provided at the critical time when a person is first offered services at a mental health clinic. During this period CTI-TS workers forge relationships that will shape the continuing use of services and enhance the potential for recovery over the subsequent course of time. The overall goal of CTI-TS is to improve the lives of those with severe mental disorders who receive community-based mental health care.

DETAILED DESCRIPTION:
Critical Time Intervention-Task Shifting (CTI-TS)is delivered by lay Community Mental Health Workers (CMHWs) and Peer Support Workers (PSWs) based in mental health outpatient service programs (MHS) and supervised by mental health professionals. These workers provide community outreach and support to engage service users, their families, primary care practitioners, peers and other community members in the recovery process.

The CTI-TS program is concerned with improving supports for people recovering from episodes of mental illness. Examples of areas where extra support may be provided include medication management, housing or crisis management, help with the family, help obtaining good services from mental health centers and primary health centers, and help developing social relationships in the community.

The program is provided by a CTI-TS team, including a community mental health worker and a peer support worker (someone who has used mental health services in the past, and has recovered). All of the CTI-TS activities will last 9 months. The evaluation of how people fare will last 18 months. The activities of CTI-TS will be in addition to the usual care provided by the subject's local health service. Usual care might include meeting with a mental health professional, meeting with a social worker, and/or obtaining prescriptions for medicine. This study will compare how people fare who have participated in the CTI-TS activities against the group of people who received only the regular services of this community mental health center. As part of the study, a trained researcher will meet with each subject for an interview at the beginning of the project, again 9 months later, and again after 18 months. These interviews will ask questions about how the subject is doing with his/her health and quality of life, and if the subject is getting help or support with problems.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age.
* No longer than 6 months since the first visit to the MHS (excluding visits that took place more than one year ago).
* Any psychotic disorder (chart diagnosis) from the following groups (ICD-10 criteria):

F20-29 including schizophrenia, delusional disorders, schizotypal disorders, acute polymorph psychotic disorders, schizoaffective disorders

F30-39 the following mood [affective] disorders with psychoses:

F30.2 Mania with psychotic symptoms F31.2 Bipolar affective disorder, current episode manic with psychotic symptoms F31.5 Bipolar affective disorder, current episode severe depression with psychotic symptoms F32.3 Severe depressive episode with psychotic symptoms F33.3 Recurrent depressive disorder, current episode severe with psychotic symptom

Exclusion Criteria:

* Under age 21 or over age 65.
* Active suicidal ideation.
* Substance Abuse or Dependence alone (may have psychotic symptoms but does not meet criteria for diagnoses included).
* Serious cognitive or other sensorial impairment which is likely to preclude reliable assessment via our interview procedures.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Camberwell Assessment of Need (CAN) | 18 months
  Used to assess the needs of people with severe mental illness.
World Health Organization Quality of Life, Short Form (WHOQOL-BREF) | 18 months
  Used to provide a quality of life measurement.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule II (WHODAS 2.0) | 18 months
  Measures level of disability
Recovery Assessment Scale (RAS) | 18 months
  Assessment tool to measure factors important to recovery
Continuity of care and course of illness | 18 months
  CONNECT, a measure of continuity of care, and the Life Chart Schedule are used.
Perceived stigma | 18 months
  Perceived Discrimination and Devaluation Scale (PDD) is used for this outcome
Self-stigma | 18 months
  Internalized stigma of mental illness (ISMI) is the measure used.
Substance use | 18 months
  ASSIST, the WHO Alcohol, Smoking and Substance Involvement Screening Test is used for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Susser, MD, DrPH, Principal Investigator — Columbia University; Graciela Rojas, MD, Principal Investigator — University of Chile; Sandro Galea, MD DrPH, Principal Investigator — Boston University; Ruben Alvarado, MD PhD, Principal Investigator — University of Chile
Locations (2):
- Federal University of Rio de Janeiro, Rio de Janeiro, Brazil
- University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang LH, Valencia E, Alvarado R, Link B, Huynh N, Nguyen K, Morita K, Saavedra M, Wong C, Galea S, Susser E. A theoretical and empirical framework for constructing culture-specific stigma instruments for Chile. Cad Saude Colet. 2013;21(1):71-79. doi: 10.1590/s1414-462x2013000100011. PMID 23990755
- [Background] Baumgartner JN, Susser E. Social integration in global mental health: what is it and how can it be measured? Epidemiol Psychiatr Sci. 2013 Mar;22(1):29-37. doi: 10.1017/S2045796012000303. Epub 2012 May 25. PMID 22794167
- [Background] Minoletti A, Galea S, Susser E. Community Mental Health Services in Latin America for People with Severe Mental Disorders. Public Health Rev. 2012;34(2):http://www.publichealthreviews.eu/show/a/116. doi: 10.1007/BF03391681. PMID 25339792
- [Background] Herman D, Opler L, Felix A, Valencia E, Wyatt RJ, Susser E. A critical time intervention with mentally ill homeless men: impact on psychiatric symptoms. J Nerv Ment Dis. 2000 Mar;188(3):135-40. doi: 10.1097/00005053-200003000-00002. PMID 10749277
- [Background] Jones K, Colson PW, Holter MC, Lin S, Valencia E, Susser E, Wyatt RJ. Cost-effectiveness of critical time intervention to reduce homelessness among persons with mental illness. Psychiatr Serv. 2003 Jun;54(6):884-90. doi: 10.1176/appi.ps.54.6.884. PMID 12773605
- [Background] Herman DB, Conover S, Gorroochurn P, Hinterland K, Hoepner L, Susser ES. Randomized trial of critical time intervention to prevent homelessness after hospital discharge. Psychiatr Serv. 2011 Jul;62(7):713-9. doi: 10.1176/ps.62.7.pss6207_0713. PMID 21724782
- [Background] Susser E, Valencia E, Conover S, Felix A, Tsai WY, Wyatt RJ. Preventing recurrent homelessness among mentally ill men: a "critical time" intervention after discharge from a shelter. Am J Public Health. 1997 Feb;87(2):256-62. doi: 10.2105/ajph.87.2.256. PMID 9103106
- [Background] Agrest M, Le PD, Yang LH, Mascayano F, Alves-Nishioka S, Dev S, Kankan T, Tapia-Munoz T, Sawyer S, Toso-Salman J, Dishy GA, Jorquera MJ, Schilling S, Pratt C, Price L, Valencia E, Conover S, Alvarado R, Susser ES. Implementing a community-based task-shifting psychosocial intervention for individuals with psychosis in Chile: Perspectives from users. Int J Soc Psychiatry. 2019 Feb;65(1):38-45. doi: 10.1177/0020764018815204. PMID 30791796
- [Background] Baumgartner JN, da Silva TF, Valencia E, Susser E. Measuring social integration in a pilot randomized controlled trial of critical time: intervention-task shifting in Latin America. Cad Saude Colet. 2012 Jan;20(4):10.1590/S1414-462X2012000400005. doi: 10.1590/S1414-462X2012000400005. PMID 24288454
- [Background] Yang L, Pratt C, Valencia E, Conover S, Fernandez R, Burrone MS, Cavalcanti MT, Lovisi G, Rojas G, Alvarado R, Galea S, Price LN, Susser E. RedeAmericas: building research capacity in young leaders for sustainable growth in community mental health services in Latin America. Glob Ment Health (Camb). 2017 Feb 14;4:e3. doi: 10.1017/gmh.2017.2. eCollection 2017. PMID 28596904
- [Background] Mascayano F, Alvarado R, Andrews HF, Jorquera MJ, Lovisi GM, Souza FM, Pratt C, Rojas G, Restrepo-Toro ME, Fader K, Gorroochurn P, Galea S, Dahl CM, Cintra J, Conover S, Burrone MS, Baumgartner JN, Rosenheck R, Schilling S, Sarucao KR, Stastny P, Tapia E, Cavalcanti MT, Valencia E, Yang LH, Susser E. Implementing the protocol of a pilot randomized controlled trial for the recovery-oriented intervention to people with psychoses in two Latin American cities. Cad Saude Publica. 2019 May 2;35(4):e00108018. doi: 10.1590/0102-311X00108018. PMID 31066775
- [Derived] Mascayano F, Alvarado R, Andrews HF, Baumgartner JN, Burrone MS, Cintra J, Conover S, Dahl CM, Fader KM, Gorroochurn P, Galea S, Jorquera MJ, Lovisi GM, Mitkiewicz de Souza F, Pratt C, Restrepo-Toro ME, Rojas G, Rodrigues Sarucao K, Rosenheck R, Schilling S, Shriver T, Stastny P, Tapia E, Cavalcanti MT, Valencia E, Yang LH, Restrepo Henao A, Martinez-Ales G, Romero Pardo V, Gomez Alemany T, Susser E. A Recovery-Oriented Intervention for People With Psychosis: A Pilot Randomized Controlled Trial. Psychiatr Serv. 2022 Nov 1;73(11):1225-1231. doi: 10.1176/appi.ps.202000843. Epub 2022 Jun 9. PMID 35678081
- See also: RedeAmericas is a National Institute of Mental Health (NIMH)-funded regional network or 'hub' for public mental health research in Latin America. — http://www.cugmhp.org/research/redeamericas/